CLINICAL TRIAL: NCT02999737
Title: Evaluating the Efficacy of Different Platelet Rich Plasma (PRP) Treatment Regimens in the Management of Androgenetic Alopecia: an Investigator-initiated, Single-center, Single-blinded, Prospective, Randomized Clinical Trial
Brief Title: Comparing Different Platelet Rich Plasma (PRP) Treatment Regimens for Management of Androgenic Alopecia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Skin Care and Laser Physicians of Beverly Hills (Other)
Collaborators: Eclipse Aesthetics, LLC (Other)
Responsible Party: Principal Investigator, Amelia K Hausauer, MD, Principal Investigator, Skin Care and Laser Physicians of Beverly Hills
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AGA-2016
Record Dates: First submitted 2016-12-19; First posted 2016-12-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Androgenetic Alopecia
Keywords: Platelet Rich Plasma; PRP; Hair loss; Alopecia; Hypotrichosis; Hair diseases
MeSH Terms: conditions — Alopecia; Hypotrichosis; Hair Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Platelet Rich Plasma for 4 sessions (Other): Autologous Platelet Rich Plasma injected in the scalp monthly x 3 then every 3 months x 1
  Interventions: Biological: Platelet Rich Plasma for 4 sessions
- Platelet rich plasma for 2 sessions (Other): Autologous Platelet Rich Plasma injected in the scalp every 3 months
  Interventions: Biological: Platelet rich plasma for 2 sessions

INTERVENTIONS:
Biological: Platelet Rich Plasma for 4 sessions — Injection of autologous platelet rich plasma into areas of alopecia on the scalp every month x 3 sessions then every 3 months x 1 session (total 4 sessions)
  Arms: Platelet Rich Plasma for 4 sessions
Biological: Platelet rich plasma for 2 sessions — Injection of autologous platelet rich plasma into areas of alopecia on the scalp every 3 months x 2 sessions (total 2 sessions)
  Arms: Platelet rich plasma for 2 sessions

SUMMARY:
The injection of autologous platelet rich plasma (PRP) is a relatively novel therapy, generating interest across a wide variety of medical specialties, such as orthopedics, dentistry, ophthalmology, and dermatology. Several recently published studies have demonstrated efficacy in treating androgenetic alopecia (aka male or female patterned hair loss), but each varies in the treatment protocol, and there is no evidence-based data to date guiding the dosing parameters of and intervals between injection sessions. We propose a single-center, single-blinded randomized pilot trial to investigate the most beneficial number and frequency ('schedule') of necessary PRP injections in men and women with androgenetic alopecia.

DETAILED DESCRIPTION:
Androgenetic alopecia is the most common form of hair loss, affecting up to 50% of men and 21 million women in the US alone. Irrespective of gender, balding is known to influence social interactions and cause substantial emotional distress, especially for those who begin losing their hair at an early age. Topical minoxidil and oral finasteride are currently the only Food and Drug Administration (FDA)-approved therapies for androgenetic alopecia in men, and oral agents are used off-label in women but are contraindicated during pregnancy and lactation. Response to these therapies varies, and they require continued use to maintain the benefits. Hair transplantation surgery is a more permanent, yet costly, solution. All of these treatments carry a risk of undesirable side effects, so there is demand for innovative new therapeutic options. Autologous platelet rich plasma (PRP) injection is a novel therapy for the treatment of patterned hair loss, but no studies to date evaluate different treatment protocols head-to-head. Hence, the purpose of this study is to compare the efficacy of two different PRP treatment schedules (frequency and number of injection sessions) in men and women with androgenetic alopecia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-65 years with AGA
* Completed and signed consent form
* Norwood Hamilton stage II-V in men or Ludwig stage I2-II1 in women
* In general good health
* Willing and able to attend all study visits
* Willing to maintain the same hair style and hair care routine as at the screening visit for the duration of the study
* Willing to have blood drawn

Exclusion Criteria:

* Younger than 18 years or older than 65 years
* Diagnosis of alopecia areata or other non-AGA forms of hair loss
* Current skin disease, cuts, or abrasions on the scalp (i.e. psoriasis, severe seborrheic dermatitis) that may limit data interpretation or put the subject at increased risk
* Scalp infection
* Malignancy, except for non-scalp nonmelanoma or melanoma skin cancers, or undergoing chemotherapy or radiation treatments
* Known history of autoimmune thyroid disease, any other thyroid disorder, or other autoimmune disorders that may interfere or increase risks associated with the study treatment
* Pregnancy, anticipated pregnancy, or breastfeeding
* Tendency to develop keloids
* History of surgical correction of hair loss on the scalp
* Use of products, devices, or medications intended to promote hair growth, except for subjects whose hair has been stable on FDA-approved therapies (i.e. oral finasteride and/or topical minoxidil) for 12 months
* Use of anti-androgenic therapies (i.e. spironolactone, flutamide, cyproterone, acetate, cimetidine) within 90 days prior to he screening visit
* Current anticoagulant therapy, except for subjects taking aspirin or other nonsteroidal anti-inflammatory drugs who are able to interrupt the medication for seven days before treatment or for subjects taking vitamin E or other over-the-counter supplements who are able to interrupt the medication for 14 days before treatment
* Hereditary or acquired hematologic/coagulation disorders including: platelet dysfunction syndrome or thrombocytopenia (count < 150,000 platelets/Ul), hypofibrinogenemia, impaired coagulation, drepanocytosis (sickle cell anemia)
* Hemodynamic instability

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-11; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Percent change in terminal hair counts | 6 months
  Evaluate the mean change in terminal hair counts (hairs/cm2) from baseline at 3 and 6 months after initial platelet rich plasma treatment

SECONDARY OUTCOMES:
Percent change in terminal hair shaft caliber | 6 months
  Evaluate the mean change in terminal hair shaft caliber (microns) from baseline at 3 and 6 months after initial platelet rich plasma treatment
Degree of hair shedding | 6 months
  Evaluate the degree of hair shedding from baseline at 3 and 6 months after initial platelet rich plasma treatment
Changes in investigator assessment of hair growth | 6 months
  Evaluate changes in the blinded investigator's overall assessment of hair growth from baseline at 3 and 6 months
Changes in subject assessment of hair growth and satisfaction | 6 months
  Evaluate changes in the subject's overall assessment of hair growth and satisfaction from baseline at 3 and 6 months
Safety and tolerability monitoring | 6 months
  Monitor for adverse effects from and tolerability of injections

CONTACTS AND LOCATIONS:
Overall Officials: Amelia K Hausauer, MD, Principal Investigator — Skincare and Laser Physicians of Beverly Hills
Locations (1):
- Skincare and Laser Physicians of Beverly Hills, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sinclair R. Male pattern androgenetic alopecia. BMJ. 1998 Sep 26;317(7162):865-9. doi: 10.1136/bmj.317.7162.865. No abstract available. PMID 9748188
- [Background] Cash TF. The psychological effects of androgenetic alopecia in men. J Am Acad Dermatol. 1992 Jun;26(6):926-31. doi: 10.1016/0190-9622(92)70134-2. PMID 1607410
- [Background] Gkini MA, Kouskoukis AE, Tripsianis G, Rigopoulos D, Kouskoukis K. Study of platelet-rich plasma injections in the treatment of androgenetic alopecia through an one-year period. J Cutan Aesthet Surg. 2014 Oct-Dec;7(4):213-9. doi: 10.4103/0974-2077.150743. PMID 25722600
- [Background] Gentile P, Garcovich S, Bielli A, Scioli MG, Orlandi A, Cervelli V. The Effect of Platelet-Rich Plasma in Hair Regrowth: A Randomized Placebo-Controlled Trial. Stem Cells Transl Med. 2015 Nov;4(11):1317-23. doi: 10.5966/sctm.2015-0107. Epub 2015 Sep 23. PMID 26400925
- [Background] Alves R, Grimalt R. Randomized Placebo-Controlled, Double-Blind, Half-Head Study to Assess the Efficacy of Platelet-Rich Plasma on the Treatment of Androgenetic Alopecia. Dermatol Surg. 2016 Apr;42(4):491-7. doi: 10.1097/DSS.0000000000000665. PMID 27035501